CLINICAL TRIAL: NCT02172196
Title: Relative Bioavailability of Both BI 10773 and Sitagliptin After Co-administration Compared to Multiple Oral Doses of BI 10773 (50 mg q.d.) Alone and Sitagliptin (100 mg q.d.) Alone in Healthy Male Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Bioavailability of BI 10773 and Sitagliptin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.27
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Sitagliptin Phosphate

ARMS (2):
- Treatment sequence ABC (Experimental): 1. Treatment A: BI 10773 once daily from day 1 to 5
  2. Treatment B: BI 10773 and sitagliptin once daily from day 1 to 5
  3. Treatment C: Sitagliptin once daily from day 1 to 5
  Interventions: Drug: BI 10773; Drug: Sitagliptin
- Treatment sequence CAB (Experimental): 1. Treatment C: Sitagliptin once daily from day 1 to 5
  2. Treatment A: BI 10773 once daily from day 1 to 5
  3. Treatment B: BI 10773 and sitagliptin once daily from day 1 to 5
  Interventions: Drug: BI 10773; Drug: Sitagliptin

INTERVENTIONS:
Drug: BI 10773
Drug: Sitagliptin

SUMMARY:
The objective was to investigate whether there was a drug-drug interaction between BI 10773 and sitagliptin when co-administered as multiple oral doses. Therefore, the relative bioavailabilities of BI 10773 and sitagliptin were determined when both drugs were given in combination compared with BI 10773 or sitagliptin given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers according to the following criteria:

  * Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age 18 to 50 years (incl.)
* BMI 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to first study drug administration
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (average consumption of more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (Torsades de pointes) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Days 1-8
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Days 1-8

SECONDARY OUTCOMES:
C24,N (concentration of analyte in plasma at 24 hours post-drug administration after administration of the Nth dose) | Days 1-8
λz,ss (terminal half-life of the analyte in plasma) | Days 1-8
t½,ss (terminal half-life of the analyte in plasma at steady state) | Days 1-8
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Days 1-8
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | Days 1-8
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | Days 1-8
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | Days 1-8
Aet1-t2,ss (amount of analyte eliminated in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
fet1-t2,ss (fraction of analyte excreted unchanged in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
CLR,ss (renal clearance of the analyte at steady state) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
UGE0-24 (Urinary glucose excretion of the analyte in urine over the time interval from time zero to 24 h) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
Abnormal findings in physical examination | Baseline and within 3-10 days after last study drug administration
Changes from baseline in vital sings (blood pressure, pulse rate) | Baseline, day 1 and within 3-10 days after last study drug administration
Changes from baseline in 12-lead ECG (electrocardiogram) | Baseline and within 3-10 days after last study drug administration
Changes from baseline in clinical laboratory tests | Baseline, day 1, 5 and within 3-10 days after last study drug administration
Incidence of adverse events | up to 28 days
Assessment of tolerability by investigator on a 4-point scale | Within 3-10 days after last study drug administration